CLINICAL TRIAL: NCT06656377
Title: Optimization of Exercise Protocol for Prediabetic Population in Postprandial State
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: DIR/KMU-EB/OE/00060; Ref No. 20-16057/NRPU/R&D/HEC (Other Grant/Funding Number: HIGHER EDUCATION COMMISSION)
Record Dates: First submitted 2024-10-14; First posted 2024-10-24 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Prediabetes; Exercise; Blood Glucose Profile; Lipid Profile; Optimization; Time
Keywords: prediabetes; Exercise; Optimization; Time; Intensity; Duration
MeSH Terms: conditions — Prediabetic State; Motor Activity

STUDY DESIGN:
Intervention Model Description: In this interventional study, we will include prediabetic patients who will undergo three sequential exercise protocols to optimize exercise timing, intensity, and duration. Each protocol is designed to explore a unique combination of these exercise parameters, allowing us to assess the effects on health outcomes relevant to prediabetes management. By using a randomized, cross-over design, participants will experience different exercise regimens, enabling us to compare the impact of each combination on glucose control, cardiovascular health, and overall metabolic function. This study aims to develop evidence-based exercise guidelines specifically tailored to prediabetic individuals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- optimizing exercise timing, intensity and duration with Prediabetes post meal (Experimental): The study is a sequential study design where a cohort of 25 will enter timing, intensity and duration protocols of exercise over 12 visits 7 days apart.
  Interventions: Behavioral: exercise intervention

INTERVENTIONS:
Behavioral: exercise intervention — A total of 25 prediabetic adults of either gender will participate in the study they will engage in exercise at intensities of 50%, 60%, 70%, or 80% of their predicted maximum heart rate (PMHR). In duration they will exercise for 15, 30, 45 and 60 minutes, and in timing protocol they will exercise at various time points after having breakfast. Blood samples were collected at four time points i.e. at fasting, pre-exercise and post-exercise at 30 and 60 minutes to measure glucose, insulin, and C-peptide levels.

SUMMARY:
The core purpose of the project is to find out optimal exercise protocol for control of hyperglycemia and insulin resistance in prediabetic. The results of the study will increase the current understandings of how exercise can be used in the most efficient manner to extract the maximum possible benefits and enhance adherence in best scientific manner possible.

DETAILED DESCRIPTION:
Participants will be selected from Peshawar and the study will be carried in accordance with the ethical code of research as per the revised (2013) declaration of Helsinki 1975. The volunteers will be recruited through posters, banners and personal contacts. The aims, objectives, purpose and procedure of the study will be explained to each participant. A written informed consent from all the participants will be taken after agreement and they will be informed about their right to leave the trial at any time if they don't want.

After selection, the recruited, participants will be asked to attend the lab for 12 visits over 6 months. On the day of experiment, patients will be received in Lab in fasting state, where baseline measurements, weight, age, BMI, W/H ratio, body composition will be determined. They will be screened for exercise fitness through PAR_Q and exercise readiness questionnaire. Detailed history of the patients (Diabetes Mellitus, medications, and economic conditions) and General Physical Examination will be carried out.

This study will be triphasic during which optimal timing of the exercise in post prandial state, optimal intensity of the exercise and optimal duration of the exercise will be quantified. For this a single cohort of 12 participants will be selected with crossover design who will attend the lab 12 times in total for all phases (04 visits for single phase). Each participant will attend the lab 12 times in total during the intervention. Each participant will be provided with one week time as wash out period.

The details of the actual visits of participants to Physiology Skill lab in detail is as under:

TIMING Protocol:

This protocol is aimed to determine the best possible time for exercise execution in postprandial state for prediabetics. During this protocol all the participants will visit the lab 04 times (7 days apart) in fasting and will be served with isocaloric breakfast (250 Kcal) after which the exercise will be started at different intervals with the following details:

Visit 1:

The participants will perform exercise 30 minutes after a standard isocaloric breakfast provided at the lab. Each exercise session will last for 40 minutes (05 minutes warm up, 05 minutes cool down) at moderate intensity (50% predicted maximum heart rate) on treadmill. Blood samples (05 ml approximately) will be taken at fasting, before exercise and 30 and 60 minutes after exercise for determination of blood glucose level, insulin, lipid profile and MicroRNAs (miR-192, miR193b).

Visit 2: - The participants will perform exercise 60 minutes after a standard isocaloric breakfast provided at the lab. Each exercise session will last for 40 minutes (05 minutes warm up, 05 minutes cool down) at moderate intensity (50% predicted maximum heart rate) on treadmill. Blood samples (05 ml approximately) will be taken at fasting, before exercise and 30 and 60 minutes after exercise for determination of blood glucose level, insulin, lipid profile and MicroRNAs (miR-192, miR193b).

Visit 3: - The participants will perform exercise 90 minutes after a standard isocaloric breakfast provided at the lab. Each exercise session will last for 40 minutes (05 minutes warm up, 05 minutes cool down) at moderate intensity (50% predicted maximum heart rate) on treadmill. Blood samples (05 ml approximately) will be taken at fasting, before exercise and 30 and 60 minutes after exercise.

Visit4: - The participants will perform exercise 120 minutes after a standard isocaloric breakfast provided at the lab. Each exercise session will last for 40 minutes (05 minutes warm up, 05 minutes cool down) at moderate intensity (50% predicted maximum heart rate) on treadmill. Blood samples (05 ml approximately) will be taken at fasting, before exercise and 30 and 60 minutes after exercise.

This protocol will provide us an optimal time for exercise in post prandial state.

Intensity Protocol:

This protocol is aimed to determine the best possible intensity of exercise in postprandial state for prediabetics. During this protocol all the participants will visit the lab 04 times (at least 2 days apart) in fasting and will be served with isocaloric breakfast (250 Kcal) after which the exercise will be started at the optimal time determined through previous protocol at different sub maximal intensities with the following details:

Visit 1:

The participants will perform exercise at 50% of predicted maximum heart rate (PMHR). Each exercise session will last for 40 minutes (05 minutes warm up, 05 minutes cool down) on treadmill. Blood samples (05 ml approximately) will be taken at fasting, before exercise and 30 and 60 minutes after exercise.

Visit 2: - The participants will perform exercise at 60% of predicted maximum heart rate (PMHR). Each exercise session will last for 40 minutes (05 minutes warm up, 05 minutes cool down) on treadmill. Blood samples (05 ml approximately) will be taken at fasting, before exercise and 30 and 60 minutes after exercise.

Visit 3: - The participants will perform exercise 70% of predicted maximum heart rate (PMHR). Each exercise session will last for 40 minutes (05 minutes warm up, 05 minutes cool down) on treadmill. Blood samples (05 ml approximately) will be taken at fasting, before exercise and 30 and 60 minutes after exercise.

Visit4: - The participants will perform exercise 80% of predicted maximum heart rate (PMHR). Each exercise session will last for 40 minutes (05 minutes warm up, 05 minutes cool down) on treadmill. Blood samples (05 ml approximately) will be taken at fasting, before exercise and 30 and 60 minutes after exercise. However, this session might need fitness of the individuals and may be omitted for some participants based on their fitness level.

Duration Protocol:

This protocol is aimed to determine the best possible duration for exercise in postprandial state for prediabetics. During this protocol all the participants will visit the lab 04 times (at least 2 days apart) in fasting and will be served with isocaloric breakfast (250 Kcal) after which the exercise will be started at the optimal time and intensity determined through previous protocols for different durations with the following details:

Visit 1:

The participants will perform exercise at optimal timing and intensity determined previously for 15 minutes excluding warm up and cool down. Blood samples (05 ml approximately) will be taken at fasting, before exercise and 30 and 60 minutes after exercise.

Visit 2: - The participants will perform exercise at optimal timing and intensity determined previously for 30 minutes excluding warm up and cool down. Blood samples (05 ml approximately) will be taken at fasting, before exercise and 30 and 60 minutes after exercise.

Visit 3: - The participants will perform exercise at optimal timing and intensity determined previously for 45 minutes excluding warm up and cool down. Blood samples (05 ml approximately) will be taken at fasting, before exercise and 30 and 60 minutes after exercise.

Visit4: - The participants will perform exercise at optimal timing and intensity determined previously for 60 minutes excluding warm up and cool down. Blood samples (05 ml approximately) will be taken at fasting, before exercise and 30 and 60 minutes after exercise.

However, this session might need fitness of the individuals and may be omitted for some participants based on their fitness level.

Analysis Procedure:

Sample analysis:

Blood glucose levels will be determined through glucometer and Insulin levels will be determined through sandwich Elisa. MicroRNAs will be extracted and then analyzed through real-time qPCR or microarray analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Prediabetic adults between 20-to-35-year age group with and without a family history of diabetes mellitus will be recruited into the study.
2. Diagnosis of prediabetes will be made through HbA1c (prediabetic range is 5·7 - 6·4%), and impaired fasting glucose (fasting plasma glucose 5·6 -6·9 mmol/L) -

Exclusion Criteria:

1. Participants with type 2 diabetes and other diseases, on lipid-lowering drugs, pregnant and lactating females or participating in some other study.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Exercise timings and Metabolic health: Targeting Blood glucose in Adults with Prediabetes post meal | 8 months
  This study aims to investigate the effects of varied exercise timing post-meal (30 min, 60 min, 90 min, and 120 minutes) on blood glucose levels. The Blood glucose levels will be measured at fasting, pre-exercise, 30 and 60 minutes post-exercise in mg/dL, using a standard glucose meter.
Exercise Timing and Metabolic health: Targeting Blood Insulin in Adults with Prediabetes post meal | 8 months
  his study aims to investigate the effects of varied exercise timing post-meal (30 min, 60 min, 90 min and 120 minutes) on Insulin levels. The Insulin levels will be measured at baseline, pre-exercise, 30 and 60 minutes post exercise, in the prediabetic population, to identify which intensity is the most effective time and improves these metabolic markers. Insulin levels will be measured using enzyme-linked immunosorbent assay (ElISA), reported in μU/mL.
Exercise timings and Metabolic health: Targeting C-peptide levels in Adults with Prediabetes post meal | 8 months
  This study aims to investigate the effects of varied exercise timing post-meal (30 minutes, 60 min, 90 min, and 120 minutes) on C-peptide levels. C-peptide levels will be assessed at fasting, pre-exercise, and 30 and 60 minutes post exercise using an enzyme-linked immunosorbent assay (ELISA) and reported in ng/mL.
Exercise timings and Metabolic health: Targeting Lipid profile levels in Adults with Prediabetes post meal | 8 months
  This study aims to investigate the effects of varied exercise timing post-meal (30 minutes, 60 min, 90 min, and 120 minutes) on Lipid profile. The lipid profile, including total cholesterol, LDL, HDL, and triglycerides, will be measured in mg/dL. Measurements will be taken at baseline and at each post-exercise interval. The outcome will determine the exercise timing that leads to the most favorable lipid profile changes.
Exercise timings and Metabolic health: Targeting MiRNA 192 expression levels in Adults with Prediabetes post meal | 8 months
  This study aims to investigate the effects of varied exercise timing post-meal (30 minutes, 60 min, 90 min, and 120 minutes) on MiRNA-192. miRNA 192 expression levels will be measured using Real-time quantitative PCR (qPCR) techniques, with results presented as relative expression values. This outcome aims to identify which exercise timing most effectively influences miRNA 192 expression.
Exercise Intensities and Metabolic health: Targeting Blood glucose levels in Adults with Prediabetes post meal | 8 months
  This study aims to investigate the effects of varied exercise intensities (50%,60%,70%, and 80%) on previously optimized meal intake time and commencement of exercise on blood glucose levels in a prediabetic population, to identify which intensity is that most effective and improves these metabolic markers. Blood glucose levels will be measured at baseline and at each post-exercise interval (30, 60, 90, and 120 minutes) in mg/dL, using a standard glucose meter.
Exercise Intensities and Metabolic health: Targeting Insulin levels in Adults with Prediabetes post meal | 8 months
  This study aims to investigate the effects of varied exercise intensities (50%,60%,70%, and 80%) on previously optimized meal intake time and commencement of exercise on insulin levels in the prediabetic population, to identify which intensity is that most effective and improves these metabolic markers. Insulin levels will be measured at the same intervals using enzyme-linked immunosorbent assay Elisa, reported in μU/mL.
Exercise Intensities and Metabolic health: Targeting C-peptide levels in Adults with Prediabetes post meal | 8 months
  This study aims to investigate the effects of varied exercise intensities (50%,60%,70%, and 80%) on previously optimized meal intake time and commencement of exercise on C-peptide levels in the prediabetic population, to identify which intensity is the most effective and improves these metabolic markers. It will be measured at the same intervals using enzyme-linked immunosorbent assay Elisa, reported in ng/mL.
Exercise Intensities and Metabolic health: Targeting Lipid Profile in Adults with Prediabetes post meal | 8 months
  This study aims to investigate the effects of varied exercise intensities (50%,60%,70%, and 80%) on previously optimized meal intake time and commencement of exercise on Lipid profile. The lipid profile, including total cholesterol, LDL, HDL, and triglycerides, will be measured in mg/dL. Measurements will be taken at baseline and at each post-exercise interval. The outcome will determine the exercise timing that leads to the most favorable lipid profile changes.
Exercise Intensities and Metabolic health: Targeting MiRNA-192 in Adults with Prediabetes post meal | 8 months
  This study aims to investigate the effects of varied exercise intensities (50%,60%,70%, and 80%) on previously optimized meal intake time and commencement of exercise on MiRNA-192. miRNA 192 expression levels will be measured using quantitative PCR (qPCR) techniques, with results presented as relative expression values. This outcome aims to identify which exercise timing most effectively influences miRNA 192 expression.
Exercise duration and Metabolic health: Targeting Blood glucose levels in Adults with Prediabetes post meal | 8 months
  This study aims to investigate the effects of varied exercise duration of exercise (15, 30, 45, and 60 minutes workout) on previously optimized time and intensity on blood glucose levels. Blood glucose levels will be measured in mg/dL, using a standard glucose meter. The goal is to determine which exercise timing results in the most significant reduction in blood glucose levels.
Exercise duration and Metabolic health: Targeting Insulin levels in Adults with Prediabetes post meal | 8 months
  This study aims to investigate the effects of varied exercise duration of exercise (15, 30, 45, and 60 minutes workout) on previously optimized time and intensity on insulin levels in a prediabetic population, to identify whichduration is the most effective and improves this metabolic marker. insulin levels will be measured at the same intervals using a chemiluminescence immunoassay, reported in μU/mL. This outcome aims to identify the optimal timing for exercise in reducing insulin levels.
Exercise duration and Metabolic health: Targeting C-peptide in Adults with Prediabetes post meal | 8 months
  This study aims to investigate the effects of varied exercise duration of exercise (15, 30, 45, and 60 minutes workout) on previously optimized time and intensity on C-peptide levels in a prediabetic population, to identify which duration is the most effective and improves this metabolic marker. C-peptide levels will be assessed at each time point using an enzyme-linked immunosorbent assay (ELISA) and reported in ng/mL. The analysis will focus on the timing of exercise that maximizes reductions in C-peptide levels.
Exercise duration and Metabolic health: Targeting Lipid Profile in Adults with Prediabetes post meal | 8 months
  This study aims to investigate the effects of varied exercise duration of exercise (15, 30, 45, and 60 minutes workout) on previously optimized time and intensity on Lipid Profile in a prediabetic population, to identify which duration is the most effective and improves thses metabolic marker. The lipid profile, including total cholesterol, LDL, HDL, and triglycerides, will be measured in mg/dL. Measurements will be taken at baseline and at each post-exercise interval. The outcome will determine the exercise timing that leads to the most favorable lipid profile changes.
Exercise duration and Metabolic health: Targeting MiRNA-192 in Adults with Prediabetes post meal | 8 months
  This study aims to investigate the effects of varied exercise duration of exercise (15, 30, 45, and 60 minutes workout) on previously optimized time and intensity on MiRNA-192 in a prediabetic population, to identify which Duration is the most effective and improves the marker. miRNA 192 expression levels will be measured using quantitative PCR (qPCR) techniques, with results presented as relative expression values. This outcome aims to identify which exercise timing most effectively influences miRNA 192 expression.

CONTACTS AND LOCATIONS:
Overall Officials: Saman Tauqir, Mphil, Principal Investigator — Khyber Medical University Peshawar, Pakistan
Locations (1):
- Khyber Medical University, Peshawar, Khyber Pukhtoon Khwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after getting approval from the principal investigator of the study, data will be kept confidential and the privacy of the data will be ensured using password-protected devices.
Supporting Information: Study Protocol
Time Frame: January 2025 to March 2025
Access Criteria: For this study, access to individual participant data (IPD) and supporting information will be controlled Who will access Primary Investigators: Members of the research team directly involved in data analysis and interpretation.
  Qualified Researchers: External researchers with relevant qualifications and interests in this field of study who meet the study's access criteria.
  Regulatory Bodies and Ethics Committees: Individuals from authorized regulatory agencies, ethics review boards, or other monitoring bodies, if required for compliance and oversight.
  What Data Will Be Accessible De-identified IPD: Anonymized individual participant data, including key variables related to the study outcomes and participant demographics.
  Supporting Documentation: This may include the study protocol, statistical analysis plan, informed consent forms, and data dictionaries.
  Summary Reports and Aggregated Results: Aggregated data or analysis summaries may be shared as part of broader research findings.

REFERENCES:
- [Background] Rynders CA, Weltman JY, Jiang B, Breton M, Patrie J, Barrett EJ, Weltman A. Effects of exercise intensity on postprandial improvement in glucose disposal and insulin sensitivity in prediabetic adults. J Clin Endocrinol Metab. 2014 Jan;99(1):220-8. doi: 10.1210/jc.2013-2687. Epub 2013 Dec 20. PMID 24243632
- [Background] Marliss EB, Vranic M. Intense exercise has unique effects on both insulin release and its roles in glucoregulation: implications for diabetes. Diabetes. 2002 Feb;51 Suppl 1:S271-83. doi: 10.2337/diabetes.51.2007.s271. PMID 11815492
- [Background] Manders RJ, Van Dijk JW, van Loon LJ. Low-intensity exercise reduces the prevalence of hyperglycemia in type 2 diabetes. Med Sci Sports Exerc. 2010 Feb;42(2):219-25. doi: 10.1249/MSS.0b013e3181b3b16d. PMID 19927038
- [Background] Irving BA, Davis CK, Brock DW, Weltman JY, Swift D, Barrett EJ, Gaesser GA, Weltman A. Effect of exercise training intensity on abdominal visceral fat and body composition. Med Sci Sports Exerc. 2008 Nov;40(11):1863-72. doi: 10.1249/MSS.0b013e3181801d40. PMID 18845966